CLINICAL TRIAL: NCT03926455
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Trial to Determine the Safety and Immunogenicity of Typhax Delivered IM
Brief Title: Safety and Immunogenicity of Typhax, a Typhoid Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Matrivax Research and Development Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Typhax-101
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Randomized, Ascending Dose
Who Masked: Participant, Investigator
Masking Description: Study vaccine will be administered by an unblinded staff member at the clinic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Typhax 0.5 mcg (Experimental): Vaccine was administered IM on Days 0 and 28 (n=9).
  Interventions: Biological: Typhax (investigational typhoid fever candidate vaccine)
- Typhax 2.5 mcg (Experimental): Vaccine was administered IM on Days 0 and 28 (n=9).
  Interventions: Biological: Typhax (investigational typhoid fever candidate vaccine)
- Typhax 10 mcg (Experimental): Vaccine was administered IM on Days 0 and 28 (n=9).
  Interventions: Biological: Typhax (investigational typhoid fever candidate vaccine)
- Typhim Vi 25 mcg (Active Comparator): Vaccine was administered IM Day 0 (n=9) followed by placebo control on Day 28
  Interventions: Biological: Placebo; Biological: Active Comparator Typhim Vi
- Placebo (saline) (Placebo Comparator): Placebo control was administered IM Days 0 and 28 ( n=9)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Typhax (investigational typhoid fever candidate vaccine)
  Arms: Typhax 0.5 mcg; Typhax 10 mcg; Typhax 2.5 mcg
Biological: Placebo — Placebo is administered to the control group on Day 0 and 28
  Arms: Placebo (saline); Typhim Vi 25 mcg
Biological: Active Comparator Typhim Vi — A single dose of commercial typhoid fever vaccine Typhim Vi is administered on Day 0, followed by placebo control on Day 28
  Arms: Typhim Vi 25 mcg

SUMMARY:
This was a randomized, double-blind, ascending dose study conducted at a single clinical research center.

DETAILED DESCRIPTION:
Healthy adult subjects aged 18 to 55 years were assigned to 3 ascending dose cohorts of Typhax (0.5, 2.5 or 10 mcg Vi antigen). Groups of 15 subjects in each dose cohort were randomized to receive Typhax, Typhim Vi (25 mcg Vi antigen) or placebo (saline) in a ratio of 3:1:1, respectively. Typhax and placebo (saline) was administered as two dose regimen (Days 0 and 28), and Typhim Vi was given as a single dose (Day 0) with matching placebo on Day 28. All doses were administered by a unblinded third-party as 0.5 mL by intramuscular (IM) injection. Safety and reactogenicity endpoints was assessed at 14 and 28 days after the first Typhax vaccination and 14 days after the second vaccination. Immunogenicity was assessed using an enzyme-linked immunosorbent assay (ELISA) to measure anti-Vi antibody serum titers on days 0, 14, 28, 42 and 180. A positive immune response (seroconversion) by ELISA is defined as at least a 4-fold increase over baseline in the Vi-specific ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women who are not pregnant or planning to become pregnant during study duration aged 18 to 55 years.
* Clinical laboratory parameters within normal laboratory limits or not found to be clinically significant by the PI

Exclusion Criteria:

* Relevant history of physical or psychiatric illness or medical disorder that required treatment.
* Known or suspected hypersensitivity to investigational product
* Immunocompromised subjects
* Previous Typhoid vaccination or elevated anti-Vi antibodies at screening
* Known history of Typhoid infection in the previous 6 months
* Positive HIV, HBsAg, or HCV screen
* Any other condition or abnormality that, in the opinion of the Investigator, may compromise the safety of the patients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited injection site and systemic events and unsolicited adverse events following vaccination with Typhax | Days 0 up to Day 56 (= 28 Days post second vaccination)
  Solicited Injection Site reactions: Pain, Tenderness, Erythema, Induration; Solicited Systemic Reactions Fever, Headache, Joint Pain, Joint Swelling, Fatigue, Myalgia, Nausea, Vomiting, Diarrhea
Number of participants reporting adverse events following vaccination with Typhax | Days 0 up to Day 210
  Adverse events are assessed at study visits by PI for seriousness, relationship to investigational product , severity and other possible etiologies
Anti-Vi IgG antibody seroconversion and geometric mean antibody titers | Day 0 - Day 14
  The immunogenicity will be measured by ELISA for anti-Vi percent seroconversion and GMTs before and at day 14 after vaccination.
Anti-Vi IgG antibody seroconversion and geometric mean antibody titers | Day 0 - Day 28
  The immunogenicity will be measured by ELISA for anti-Vi percent seroconversion and GMTs before and at day 28 after vaccination.
Anti-Vi IgG antibody seroconversion and geometric mean antibody titers | Day 0 - Day 42
  The immunogenicity will be measured by ELISA for anti-Vi percent seroconversion and GMTs before and at day 42.
Anti-Vi IgG antibody seroconversion and geometric mean antibody titers | Day 0 - Day 180.
  The immunogenicity will be measured by ELISA for anti-Vi percent seroconversion and GMTs before and at day 180.

SECONDARY OUTCOMES:
Vi-specific B-cell ELISPOT responses | Days 0 through 38
  Immunogenicity was evaluated by comparing the number of Vi-specific B-cells by ELISPOT in PBMC samples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cartee RT, Thanawastien A, Griffin Iv TJ, Mekalanos JJ, Bart S, Killeen KP. A phase 1 randomized safety, reactogenicity, and immunogenicity study of Typhax: A novel protein capsular matrix vaccine candidate for the prevention of typhoid fever. PLoS Negl Trop Dis. 2020 Jan 6;14(1):e0007912. doi: 10.1371/journal.pntd.0007912. eCollection 2020 Jan. PMID 31905228